CLINICAL TRIAL: NCT03886194
Title: Comparative Study of Interventional and Systemic Thrombolysis in Patients With High-risk and High-risk Pulmonary Embolism
Brief Title: Thrombolytic and Interventional Treatment of Pulmonary Embolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2018-023
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrombolytic group (Active Comparator): Thrombolytic group: urokinase 20,000 units / kg body weight, 2 hours intravenous drip; or rtPA 50mg, 2 hours intravenous drip
  Interventions: Procedure: interventional treatment in pulmonary
- Interventional treatment group (Experimental): Interventional treatment group: intracavitary catheter contact thrombolysis (urokinase 500,000 u 5 minute pulse Give), catheter thromboembolism, thrombus aspiration and mechanical thrombectomy.
  Interventions: Procedure: interventional treatment in pulmonary

INTERVENTIONS:
Procedure: interventional treatment in pulmonary — Thrombolytic group: urokinase 20,000 units / kg body weight, 2 hours intravenous drip; or rtPA 50mg, 2 hours intravenous drip; and interventional treatment group: intracavitary catheter contact thrombolysis (urokinase 500,000 u 5 minute pulse Give), catheter thromboembolism, thrombus aspiration and mechanical thrombectomy.

SUMMARY:
Pulmonary embolism (PE) is a pulmonary vascular disease that seriously endangers human health. It has the characteristics of high morbidity, high mortality, high misdiagnosis rate and low detection rate. The mortality rate in March is about 10%. The high-risk and high-risk PE mortality rate is greater than 15%. Chronic thromboembolic pulmonary hypertension (CTEPH) is a serious sequelae after PE, with a poor prognosis and expensive treatment. Systemic thrombolysis is the preferred treatment for acute high-risk pulmonary embolism, which can reduce mortality, but the incidence of major bleeding is increased by 5 times and hemorrhagic stroke is increased by 10 times. Recent studies have concluded that interventional therapy is a viable approach with a high success rate, effective improvement of clinical outcomes, and minimization of major bleeding risks. However, there is no good prospective study of interventional therapy compared with systemic thrombolytic therapy. This study was enrolled in the diagnosis of high-risk and high-risk PE patients, randomized to the system of thrombolytic therapy or interventional therapy (including pulmonary artery catheter contact thrombolysis, catheter thrombectomy, thrombus aspiration and mechanical thrombectomy, etc.) Symptoms improved during surgery, right heart condition, mortality and complications, and were followed up to December to observe PE recurrence CETPH, survival and cardiopulmonary function. In order to provide new evidence for the treatment of fatal pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Han population with age greater than or equal to 14 years old and less than or equal to 85 years;
* Signed informed consent;
* confirmed initial acute pulmonary embolism, within 2 weeks of disease, pulmonary embolism confirmed methods include: CTA/DSA/pulmonary ventilation Imaging: confirmed as at least 1 trunk pulmonary artery or proximal low lobe artery filling defect;
* risk stratification for intermediate high-risk or high-risk pulmonary embolism: 2014ESC stratified definition of high-risk and high-risk: high-risk PE: hemodynamics Obstruction, systolic blood pressure <90mmHg, greater than 15 minutes; medium and high risk PE: right ventricular dysfunction imaging findings (RV / LV ≥ 0.9) and myocardial damage indicators positive (TNT > 0.1 ng / ml);
* blood flow at admission The kinetics are stable.

Exclusion Criteria:

* patients with mental illness can not cooperate with the completion of the study; -CTPA / DSA contraindications patients;
* any contraindications listed in the instructions for treatment of the drug involved in the study;
* diseases associated with coagulopathy leading to the risk of clinically relevant bleeding;
* There are active bleeding or high risk of bleeding in patients with anticoagulant thrombolysis contraindications;
* creatinine clearance rate <30 mL / min;
* life expectancy ≤ 6 months;
* childbearing age or pregnancy, lactation period without appropriate contraceptive measures Subjects;
* participated in any other drug or medical device study within 30 days prior to randomization;
* cases that the investigator considered unsuitable for participation in the trial.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-18 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Right heart load | 30 days
  RV/LV (thoracic enhanced CT/cardiac ultrasound),pulmonary artery pressure (catheter/cardiac ultrasound),troponin T, NT-proBNP, 6-minute walk test
death within 30 days | 30 days
  number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Zhang, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No